CLINICAL TRIAL: NCT02759575
Title: A Phase I/II Study of Chemo Radiation Plus the Anti-Programmed Death-1 (Anti-PD-1) Antibody, Pembrolizumab (MK-3475) for Locally Advanced Laryngeal Squamous Cell Carcinoma
Brief Title: A Study of Chemoradiation Plus Pembrolizumab for Locally Advanced Laryngeal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinita Takiar (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Vinita Takiar, Assistant Professor of Radiation Oncology, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HN-15-02
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab every 3 weeks in combination with 7 weeks of radiation therapy and every 3 week cisplatin
  Interventions: Drug: Pembrolizumab; Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — 200mg every 3 weeks starting 3 weeks prior to chemoradiotherapy. Maximum of 4 doses
  Other Names: Keytruda
Radiation: Radiation Therapy — 70 Gy in 35 fractions over 7 weeks
Drug: Cisplatin — 100 mg/m2 every 3 weeks starting on day 1 of chemoradiotherapy. Maximum of 3 doses.
  Other Names: Platinol

SUMMARY:
The purpose of this research study is to test the safety and the benefit of adding pembrolizumab (a therapy that activates the immune system to fight cancer) to standard of care treatment for larynx cancer. The standard of care treatment will include chemotherapy and radiation for 7 weeks.

DETAILED DESCRIPTION:
This study is an open label, single arm study which will enroll patients with locally advanced squamous cell carcinomas of the larynx. Positive tumor PDL1 expression by IHC will not be required for enrollment.

All patients with receive Pembrolizumab and cisplatin in combination with radiation. Pembrolizumab 200 mg flat dose given Q21 days will begin 3 weeks prior to initiation of chemoradiation and continued through the 21-day cycle until completion of chemoradiation. Cisplatin will be given 100 mg/m2 every 21 days during radiation as per standard of care.

Pembrolizumab has well defined toxicities as single agent and has non-overlapping mechanisms of action with cisplatin and radiation. The safety of these agents used in combination has not been previously described, therefore the study will begin with a safety run-in phase 1 followed by the phase II design. See statistical section for details.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven, previously untreated stage III or IV squamous cell carcinoma of the larynx, Primary tumor stage (T2, T3) and nodal stage (N0, N1, N2, N3).
* Measurable disease based on RECIST 1.1.
* Performance status 0 or 1 on Eastern Cooperative Oncology Group Performance Scale.
* Anticipated survival minimum of 12 months.
* Adequate labs

Exclusion Criteria:

* Patients with T1 primary tumor or T4 large volume tumor that has resulted in larynx dysfunction at baseline (for example tumor largely penetrating into base of tongue and resulting in inability to swallow at baseline)
* Prior radiation therapy to the larynx area or involved neck.
* Distant metastasis
* Known history of active tuberculosis (TB), autoimmune disease, pneumonitis, infection, HIV, Hepatitis B, or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinita Takiar, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Frankart AJ, Sadraei NH, Huth B, Redmond KP, Barrett WL, Kurtzweil N, Riaz MK, Wise-Draper T, Rodriguez CP, Adelstein DJ, Takiar V. A phase I/II trial of concurrent immunotherapy with chemoradiation in locally advanced larynx cancer. Laryngoscope Investig Otolaryngol. 2022 Mar 17;7(2):437-443. doi: 10.1002/lio2.780. eCollection 2022 Apr. PMID 35434343

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 54 [37 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Grade 3 or 4 Adverse Events as Assessed by CTCAE V4.0
Description: Greater than 2 grade 3 or 4 adverse events that are definitely, probably or possibly related to the pembrolizumab in the first cohort of 6 participants
Time Frame: 30 days following completion of treatment for the first 6 participants
Population: These are the first six participants that completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 6
Participants | 2

2. Primary Outcome: Laryngectomy-free Survival in Locally Advanced Laryngeal Squamous Cell Carcinoma
Description: This is the number of subjects that are laryngectomy-free at 18 months.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Laryngectomy-free Survival in Locally Advanced Laryngeal Squamous Cell Carcinoma
Description: This is the number of subjects that are laryngectomy-free at 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 9
Participants | 9

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=9)
Metabolism and nutrition disorders - Other- Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (3) — One of the events resulted in death unrelated to study participation, due to subject's compliance to diabetes treatment.
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Acute Kidney Disease (Renal and urinary disorders) | 1 (1)
Failure to Thrive (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=9)
Acute Kidney Injury (Renal and urinary disorders) | 4 (6)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Anxiety (Psychiatric disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Investigations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Dermatitis radiation (Injury, poisoning and procedural complications) | 9 (12)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 8 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 8 (15)
Dysphagia (Gastrointestinal disorders) | 7 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 8 (15)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Increased Mucus Production (General disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 2 (2)
Lymphedema (Vascular disorders) | 3 (4)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 4 (8)
Neutrophil count decreased (Investigations) | 2 (2)
Pain (General disorders) | 2 (3)
Platelet count decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Throat swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Investigations) | 6 (14)
White blood cell decreased (Investigations) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Tenderness (around feeding tube) (Injury, poisoning and procedural complications) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Localized edema (General disorders) | 2 (3)
Lymphocyte count decreased (Investigations) | 2 (3)
Mucosal infection (Infections and infestations) | 2 (2)
Sensitive fingertips (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Two white spots on ventricular fold (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intermittent lightheadedness (Nervous system disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Salivary duct inflammation (Gastrointestinal disorders) | 5 (5)
Sepsis (Infections and infestations) | 1 (1)
Dry skin of lower lip (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Stoma site infection (Infections and infestations) | 2 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02759575/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT02759575/ICF_001.pdf